CLINICAL TRIAL: NCT06974383
Title: Development and Validation of Virtual Laparoscopic Hiatal Hernia Simulator (VLaHHS)
Brief Title: Development and Validation of Virtual Laparoscopic Hiatal Hernia Simulator
Acronym: (VLaHHS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Ganesh Sankaranarayanan, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU-2021-0151; 1R01EB025247-01A1 (NIH)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Predictive Validity of VLaHHS
Keywords: Virtual Laparoscopic Hiatal Hernia Simulator (VLaHHS); GS Residents

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 2 groups - simulation group & Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Simulation Group) (Experimental): Training with VLaHHS. Before the testing session begins, all participants will receive a guided, hands-on orientation to the task that is being tested. They will then take a pre-test in which they will be asked to perform the task once to mark their baseline performance (i.e. initialize their learner profile).
  Interventions: Other: Training with Virtual Laparoscopic Hiatal Hernia Simulator (VLaHHS)
- Group 2 (Control Group) (No Intervention): No training with VLaHHS. Before the testing session begins, all participants will receive a guided, hands-on orientation to the task that is being tested. They will then take a pre-test in which they will be asked to perform the task once to mark their baseline performance (i.e. initialize their learner profile). They will continue with their normal residency training but will not participate in VLaHHS training at all.

INTERVENTIONS:
Other: Training with Virtual Laparoscopic Hiatal Hernia Simulator (VLaHHS) — For the training phase, participants in Group 1 will perform the tasks on VLaHHS for an hour a day for a maximum of 15 sessions over 3 weeks.
  Arms: Group 1 (Simulation Group)

SUMMARY:
The goal of this study is to establish the face, content, discriminant and predictive validity of the Virtual Laparoscopic Hiatal Hernia Simulator (VLaHHS). The study population includes GS residents. The goal of developing scenarios for the simulator will be accomplished first and establishing the validity of the VLaHHS will be conducted in three phases after that:

1. Needs assessment survey of current practices in laparoscopic hiatal hernia repair

a. Development of scenarios and metrics for the VLaHHS b. Assessment of validity of metrics developed for VLaHHS

3) Assessment of validity of VLaHHS

1. Phase I - Face and content Validity Assessment of VLaHHS
2. Phase II - Discriminant Validity Assessment of VLaHHS
3. Phase III - Learning Curve, Retention and Transfer Assessment (predictive validity) of VLaHHS

Part 3- Phase III of this study is the interventional portion while rest of the parts and phases do not involve an intervention. The goal of this phase of the study is to establish the learning curve and predictive validity of the VLaHHS.

The hypothesis is that the subject trained in VLaHHS will improve their skills compared to control with no training and show better transfer of skills on to an actual procedure.

DETAILED DESCRIPTION:
The learning curve of VLaHHS will be established by training subjects in the task over extended period until they reach a plateau. The predictive validity will be established by comparing the training group with a control group with no training by testing their skills on a simulated surgical task using a crural repair silicone model and porcine fundoplication model.

The experimental design is a between-subjects design with two groups to which participants will be randomly assigned: (1) Group 1 (Simulation Group): training with VLaHHS, (2) Group 2 (Control Group): no training. Two separate tasks ((1) Crural closure and (2) Fundoplication ) of VLaHHS will be tested separately (10 subjects per task). Before the testing session begins, all participants will receive a guided, hands-on orientation to the task that is being tested. They will then take a pre-test in which they will be asked to perform the task once to mark their baseline performance (i.e. initialize their learner profile). For the training phase, participants in Group 1 will perform the tasks on VLaHHS for an hour a day for a maximum of no more than three weeks (3 weeks' x 5 days = 15 sessions). In each session of no more than an hour, subjects will repeat the task five times.

Participants in Group 2 will continue with their normal residency training but will not participate in VLaHHS training at all.

Two aspects of learning will then be assessed post-training: skill learning and transfer-of-training. For the Simulation Group, skill learning will be measured immediately following training (post-test) and again after two weeks to measure retention. For the Control Group, skill learning will be measured four weeks after orientation and again two weeks later to measure retention. Finally, immediately after post-test, transfer-of-training will be assessed using simulated crural repair or fundoplication model. The transfer study will be conducted either at the UTSW Simulation Center or at the Artificial Intelligence and Medical Simulation (AIMS) Lab in south campus.

Dependent measures for learning curve and retention will be the score computed from completion time and errors on the VLaHHS and the workload assessment measured using the NASA-TLX questionnaire after each session. For the transfer task, Subjects performance on the crural repair and fundoplication task will be video recorded and evaluated by a minimum of three experts using Global Assessment Tools for Intraoperative Laparoscopic Skills (GOALS) subjective evaluation method (See Appendix AIII).

The videotaping will focus only on subjects hand and any Identifying information such as subjects face will not be captured.

ELIGIBILITY:
Inclusion Criteria:

* General Surgery (GS) residents

Exclusion Criteria:

* Residents other than GS
* Participants who are not residents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Skill level in participants as assessed by completion time | Baseline (at pre-test)
  Dependent measures for learning curve will be assessed by completion time.
Skill level in participants assessed by errors on the VLaHHS | Baseline (at pre-test)
  Dependent measures for learning curve will be assessed by errors on the VLaHHS
Skill level in participants assessed by NASA-TLX questionnaire | Baseline (at pre-test)
  Dependent measures for learning curve will be measured using the NASA-TLX questionnaire. The NASA Task Load Index (NASA-TLX) is a tool to subjectively assess cognitive and emotional load during a simulation. Students rate six dimensions: mental and physical demands, time pressure, performance, effort, and frustration. Each dimension is assessed on a scale of 0-10, where a higher value indicates a higher burden. The NASA-TLX total score can be calculated as the average of all dimensions or using weighted scoring.
Skill level in participants as assessed by completion time | Immediately post test
  Dependent measures for learning curve will be assessed by completion time.
Skill level in participants assessed by errors on the VLaHHS | Immediately post test
  Dependent measures for learning curve will be assessed by errors on the VLaHHS
Skill level in participants assessed by NASA-TLX questionnaire | Immediately post test
  Dependent measures for learning curve will be measured using the NASA-TLX questionnaire. The NASA Task Load Index (NASA-TLX) is a tool to subjectively assess cognitive and emotional load during a simulation. Students rate six dimensions: mental and physical demands, time pressure, performance, effort, and frustration. Each dimension is assessed on a scale of 0-100, where a higher value indicates a higher burden. The NASA-TLX total score can be calculated as the average of all dimensions or using weighted scoring.
Skill retention in participants as assessed by completion time | 2 weeks after post test
  Dependent measures will be assessed by completion time.
Skill retention in participants as assessed by errors on the VLaHHS | 2 weeks after post test
  Dependent measures will be assessed by errors on the VLaHHS
Skill retention in participants as assessed by NASA-TLX questionnaire | 2 weeks after post test
  Dependent measures will be assessed by NASA-TLX questionnaire. The NASA Task Load Index (NASA-TLX) is a tool to subjectively assess cognitive and emotional load during a simulation. Students rate six dimensions: mental and physical demands, time pressure, performance, effort, and frustration. Each dimension is assessed on a scale of 0-100, where a higher value indicates a higher burden. The NASA-TLX total score can be calculated as the average of all dimensions or using weighted scoring.
Transfer of skill in participants as assessed by GOALS | Immediately post test
  This measure will be assessed using Global Assessment Tools for Intraoperative Laparoscopic Skills (GOALS). It's a 5-item global rating scale that evaluates performance in areas like depth perception, bimanual dexterity, efficiency, tissue handling, and autonomy. Possible scores in each domain will range from 1-5 and total range combining each domain will be 5-25 with higher score indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Sankaranarayanan, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No